CLINICAL TRIAL: NCT00003974
Title: An Evaluation of the Immunological Parameters Associated With a Skin-Test and Immunization of Lung and Mesothelioma Cancer Patients With Autologous Lung Tumor Associated Antigen: Characterization of the Patients' Cytolytic and Helper T Cell Reactivity for Identification of the Specific Antigen(s): A Pilot Study
Brief Title: Vaccine Therapy in Treating Patients With Stage I, Stage II, or Stage IIIA Non-small Cell Lung Cancer or With Stage I or Stage II Mesothelioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Timothy M. Anderson, MD, Roswell Park Cancer Institute
Purpose: Treatment
Other Study IDs: CDR0000067177; RPCI-DS-96-25
Record Dates: First submitted 1999-11-01; First posted 2004-08-20 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Lung Cancer; Malignant Mesothelioma
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; localized malignant mesothelioma; stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Mesothelioma, Malignant; Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: lung tumor associated antigen
Drug: DetoxPC
Drug: chemotherapy
Drug: cyclophosphamide

SUMMARY:
RATIONALE: Vaccines made from a person's tumor may help the body build an immune response to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy in treating patients who have undergone surgery to remove stage I, stage II, or stage IIIA non-small cell lung cancer or stage I or stage II mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Define the immunological parameters of cytolytic T cell and T helper cell activity associated with skin testing and vaccination with autologous lung tumor associated antigen and detoxPC in patients with curatively resected stage I, II, or IIIA non-small cell lung cancer (NSCLC) or stage I or II mesothelioma. II. Evaluate any responses associated with an enhanced antitumor immune status in this patient population with this treatment regimen.

OUTLINE: Patients undergo delayed type hypersensitivity skin testing with autologous tumor associated antigen (TAA) and memory antigens (i.e., Monilia, PPD, and Trichophyton) intradermally at 1-4 weeks following surgical tumor resection. At week 4-9, patients receive low dose cyclophosphamide IV once. At 3 days following chemotherapy, patients receive autologous TAA with DetoxPC intradermally for up to 3 doses over 4 weeks. At 2-3 weeks following vaccination, patients undergo repeat skin testing. At week 6-12, patients with a positive skin test undergo biopsy of the skin test/vaccination site followed by leukapheresis at week 12-20 if T cells exhibit active antitumor reactivity. Patients with stable or regressive disease receive additional vaccination courses at week 20 and thereafter. Patients are followed for 5 years.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven primary stage I (T2, N0), II, or IIIA non-small cell lung cancer (NSCLC) curatively resected by pneumonectomy, lobectomy, or wedge resection OR Stage I or II mesothelioma Measurable disease Lesions must be at least 3 cm in diameter

PATIENT CHARACTERISTICS: Age: 20 to 70 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No other malignancy except nonmelanoma skin cancer No history of severe allergies No history of autoimmune disease Not pregnant

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: No concurrent glucocorticoids Radiotherapy: Not specified Surgery: See Disease Characteristics Other: No concurrent nonsteroidal antiinflammatory drugs

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1997-08; Primary Completion 1998-06 (Actual); Study Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M. Anderson, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States